CLINICAL TRIAL: NCT01699919
Title: Effect of Perioperative Systemic Lignocaine on Postoperative Pain in Patients Undergoing Elective Open Abdominal Surgeries- a Double Blinded Randomized Control Trial
Brief Title: A Study to Assess Analgesic Efficacy of Intravenous Lignocaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Principal Investigator, Dr.P.Sridhar, Junior resident, Department of Surgery, Principal investigator, Jawaharlal Institute of Postgraduate Medical Education & Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEC No. : EC/2011/2/24
Record Dates: First submitted 2012-09-26; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting; Postoperative Ileus
Keywords: perioperative lignocaine infusion; elective open abdominal surgeries; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous lignocaine (Active Comparator): Intravenous lignocaine will be given as a bolus of 1.5mg/kg at the time of intubation followed by an infusion at a rate of 1.5mg/kg/hr throughout surgery and till one hour post surgery.
  Interventions: Drug: Intravenous lignocaine
- normal saline (Placebo Comparator): Normal saline will be given as a bolus at the time of intubation and saline infusion given to patients in the control group during the surgery and till one hour post surgery.
  Interventions: Drug: Intravenous lignocaine

INTERVENTIONS:
Drug: Intravenous lignocaine — Intravenous lignocaine infusion is given in intraoperative period and till one hour post surgery.
  Other Names: Lidocaine, Xylocard

SUMMARY:
The primary objectives of this study are to analyse the effect of perioperative systemic infusion of lignocaine on postoperative pain, postoperative nausea and vomiting and perioperative levels of inflammatory mediators in patients undergoing elective open abdominal surgeries.

The secondary parameters which will be observed during the study are the time to passage of flatus and stools postoperatively.

DETAILED DESCRIPTION:
Patients will be randomized into two groups- A and B, to receive an intravenous infusion of lignocaine or saline,respectively, as a bolus of 1.5mg/kg at the time of intubation followed by an infusion at a rate of 1.5mg/kg/hr continued throughout the surgery and till one hour postop. Postoperative analgesia will be provided through Patient Controlled Analgesia (PCA) pump providing morphine. Postoperative pain scores will be noted at immediate postoperative and at 6, 18, 24 hours post surgery. The number of PCA demands and cumulative morphine consumption till 24 hours post surgery will be noted. The incidence of postoperative nausea and vomiting is recorded. The time to first passage of flatus and stools postoperatively will be noted. Levels of total leukocyte count, c-reactive protein (CRP) and interleukin-6(IL-6) will be noted in preoperative, immediate post operative and 24 hours post surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years of age
* undergoing elective open abdominal surgeries
* belonging to the American Society of Anaesthesiologists (ASA)status I,II,III

Exclusion Criteria:

* patients sensitive to lignocaine,
* patients suffering from cardiovascular diseases or with preoperative changes on electrocardiogram
* patients on beta blocker drugs
* patients on opioid drugs for prolonged period
* patients with functional bowel disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
postoperative pain scores using visual analogue scale | till 24 hours post surgery
  Postoperative pain scores are assessed in the patients using a visual analogue scale in the first 24 hours post surgery

SECONDARY OUTCOMES:
Number of patient controlled analgesia demands | Till 24 hours post surgery
  The total number of times the patient presses the demand button of PCA pump are noted.
Total amount of morphine consumed | till 24 hours post surgery
  The total morphine consumption till 24 hours post surgery is noted.

OTHER OUTCOMES:
Perioperative levels of inflammatory mediators | in preoperative period, immediate post op and 24 hours post surgery
  Blood samples will be collected for the analysis of total leukocyte count, C-reactive protein and Interleukin-6 levels in the preoperative period, immediate postoperative and at 24 hours post surgery.
time of passage of flatus and stools postoperatively | till postoperative day 7
  Postoperative bowel function recovery will be assessed by noting the time of first passage of flatus and stools postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: parnandi sridhar, MBBS, Principal Investigator — Junior resident,JAWAHARLAL INSTITUTE OF POSTGRADUATE MEDICAL EDUCATION AND RESEARCH, PUDUCHERRY, INDIA
Locations (1):
- Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry, Puducherry, India

REFERENCES:
- [Background] Cassuto J, Wallin G, Hogstrom S, Faxen A, Rimback G. Inhibition of postoperative pain by continuous low-dose intravenous infusion of lidocaine. Anesth Analg. 1985 Oct;64(10):971-4. PMID 3898920
- [Background] Groudine SB, Fisher HA, Kaufman RP Jr, Patel MK, Wilkins LJ, Mehta SA, Lumb PD. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesth Analg. 1998 Feb;86(2):235-9. doi: 10.1097/00000539-199802000-00003. PMID 9459225